CLINICAL TRIAL: NCT04654637
Title: Department of Nursing, Tzu Chi University, Hualien, Taiwan
Brief Title: Multiple Interactive With Nutrition and Exercise Strategies in Frailty Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Chun Hou Huang, Assistance Professor, Tzu Chi University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: TCU-CHHuang
Record Dates: First submitted 2020-11-25; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Arm A: fix model of cycle exercise(online supervise) and routine nutrition consult Arm B: fix model of cycle exercise(online supervise) and online nutrition consult Arm C: individualize cycle exercise(online supervise) and routine nutrition consult Arm D: individualize cycle exercise(online supervise) and online nutrition consult
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): fix model of cycle exercise(online supervise) and routine nutrition consult
  Interventions: Behavioral: Nutrition and Exercise Strategies
- Arm B (Experimental): fix model of cycle exercise(online supervise) and online nutrition consult
  Interventions: Behavioral: Nutrition and Exercise Strategies
- Arm C (Experimental): individualize cycle exercise(online supervise) and routine nutrition consult
  Interventions: Behavioral: Nutrition and Exercise Strategies
- Arm D (Experimental): individualize cycle exercise(online supervise) and online nutrition consult
  Interventions: Behavioral: Nutrition and Exercise Strategies

INTERVENTIONS:
Behavioral: Nutrition and Exercise Strategies — Multiple Interactive with Nutrition and Exercise Strategies

SUMMARY:
Due to the changes in lifestyle caused by the COVID-19, it is a priority to provide multi-interactive digital platforms and social media for nutrition and exercise programs for cancer patients. A two-year serial program uses mixed study methods of longitudinal combined experimental study. We will investigate cancer frailty's current situation and track the frailty trends after cancer patients received different treatments. We will also invite experts to develop multi-interactive digital platforms of nutrition and performance-based tailored circuit training programs according to the cancer frailty survey. We will recruit 20-85 years of newly diagnosed or first-time recurrence cancer patients and stratified randomization assigned to evaluate nutrition and physical exercise intervention effectiveness. The measure indicators were treatment-related adverse events, nutritional status, frailty status, survival rate, and life quality.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 20-85 years with histological confirmation malignancy.
* Requiring treatment by surgery, chemotherapy, hormonotherapy, radiotherapy, or targeted therapy with a curative intention as estimated by oncologists.
* First diagnosed or recurrence of head and neck cancer, esophageal cancer, colon/rectum cancer, lung cancer, AML, ALL, lymphoma, multiple myeloma.

Exclusion Criteria:

* Non-head and neck cancer, esophageal cancer, colon/rectum cancer, lung cancer, AML, ALL, lymphoma, multiple myeloma with first diagnosis or recurrence patients.
* Eastern Cooperative Oncology Group test score>2.
* Serious psychiatric or cognitive problems, and functional disability leading to a total inability to walk.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Frailty trend | After treatment three-month
  After treatment frailty condition

SECONDARY OUTCOMES:
Treatment-related adverse events | After treatment one month
  CTCAE or Clavien-Dindo classification

OTHER OUTCOMES:
Survival | The OS was calculated from the date of diagnosis to the date of death or was censored at the date of the last follow-up (3 years from diagnosed) for surviving patients.
  from diagnosed to the dead date

CONTACTS AND LOCATIONS:
Locations (1):
- Tzu Chi University, Hualien City, Taiwan